CLINICAL TRIAL: NCT01901224
Title: Metformin, Muscle Energetics, and Vascular Function in Older Adults With Peripheral Artery Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: study was not funded
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Mark Alan Creager, MD, Mark A. Creager, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013P001042
Record Dates: First submitted 2013-07-12; First posted 2013-07-17 (Estimated); Results first posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Metformin 1000 mg (Experimental): metformin 1000 mg twice daily: In order to avoid gastrointestinal side effects, the starting dose of metformin will be 500 mg twice daily. After one week, the dose will be increased to 1000 mg twice daily (as two 500 mg tablets twice daily). Subjects will be instructed to take medications with breakfast and with dinner.
  Interventions: Drug: Metformin 1000 mg
- Control (Placebo Comparator): placebo twice daily: In order to maintain blinding during the titration period, individuals randomized to placebo will receive one placebo tablet twice daily for one week, followed by an increase to 2 placebo tablets twice daily. Subjects will be instructed to take medications with breakfast and with dinner.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin 1000 mg
  Arms: Metformin 1000 mg
Drug: Placebo
  Arms: Control

SUMMARY:
The investigators are doing this research study to find out if taking Metformin improves walking ability in patients with peripheral arterial disease (PAD). In PAD the arteries (blood vessels) in the legs are narrowed because of the build up of plaque. The leg muscle can hurt in patients with PAD and this is usually described as a cramp or tiredness. This pain is called intermittent claudication. Metformin is an FDA approved medication for the treatment of diabetes. The investigators believe that Metformin may help your leg muscles work better.

The investigators will enroll up to 100 subjects in order to find 60 subjects with PAD at Brigham and Women's Hospital (BWH).

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is a manifestation of atherosclerosis that affects more than 7 million adults in the US. The prevalence of PAD increases with age and is estimated to be 15 20% among individuals 65 years of age and older. Patients with PAD have limited functional capacity; they walk more slowly and have less walking endurance than persons who do not have PAD, irrespective of whether they have classic symptoms of intermittent claudication or critical limb ischemia. This functional impairment adversely affects quality of life. Although flow limitation due to atherosclerotic stenosis is necessary for the development of symptoms in PAD, the lack of correlation between walking capacity and the degree of hemodynamic compromise raises the possibility that alternative mechanisms contribute to functional limitations in these patients. Putative mechanisms include inadequate skeletal muscle glucose uptake, altered skeletal muscle energetics, and impaired vasomotor tone and nutrient delivery mediated by endothelial dysfunction. Metformin, via AMPactivated protein kinase (AMPK)-dependent and independent mechanisms, can favorably affect skeletal muscle metabolic functions including glucose uptake, fatty acid oxidation, mitochondrial function, and consequently cellular energetics, and it also may have a direct salutary effect on vascular function via regulation of nitric oxide synthase. It is intriguing, therefore, to consider the possibility that metformin would improve skeletal muscle metabolic and vascular function in older patients with PAD and translate into functional benefits. Accordingly, the investigators seek to elucidate molecular mechanisms through which metformin affects skeletal muscle energetics and hypothesize that metformin will lead to advantageous metabolic, vascular, and physical functional changes in older patients with PAD.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or greater
* Intermittent claudication for 6 months or greater
* Maximal walk time between 1-20 minutes on all ETTs
* Resting ABI ≤ 0.9 in index leg at baseline
* ABI falls ≥ 20% in index leg 1 minute post baseline ETT
* MWT variability < 20%

Exclusion Criteria:

* Type 1 or Type 2 Diabetes
* Limb-threatening ischemia (rest pain, ulceration, gangrene)
* Peripheral vascular surgery or PCI within 6 months
* MI or CABG within 6 months
* Carotid endarterectomy (CEA) within 6 months
* Cerebrovascular accident or TIA within 6 months
* Uncontrolled hypertension (SBP > 140 mmHg, DBP >90 mmHg)
* Pentoxifylline/Cilostazol added/changed within 3 months
* HMG-CoA reductase inhibitor added/changed within 3 months
* Exercise limitations other than claudication (heart failure, angina, COPD, arthritis, neuropathy, etc.)
* Serum creatinine ≥ 1.5 mg/dL
* Pregnant or plans to become pregnant
* 2 hour Oral Glucose Tolerance Test (OGTT) > 200 mg/dL

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Creager, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization blind was never broken, so only overall study participant flow is available.
Groups:
- Overall Study: Overall Study (Metformin and Placebo arms combined)
Period: Overall Study
Arm/Group | Overall Study
Started | 2
Completed | 0
Not Completed | 2
Not completed — study was not funded and terminated | 2

BASELINE CHARACTERISTICS:
Population: Randomization blind was never broken, so only overall study participant baseline measures are available.
Arm/Group | Overall Study
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.5 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in PCr Recovery Time
Description: PCr recovery time, measured in seconds, is a measure of skeletal muscle metabolic function. PCr is a transport molecule and reservoir of high-energy phosphate bonds, which is important for cellular energetics. Phosphocreatine regeneration depends upon the skeletal muscle mitochondrial cells capacity for oxidative phosphorylation. We will measure PCr recovery time at baseline and after 12 weeks of treatment with metformin or placebo as an in vivo measure of mitochondrial function. Higher Pcr relative to P(i) during recovery is better and shorter recovery times are better.
Time Frame: baseline, 12 weeks
Population: Study was not funded and was terminated prematurely. Randomization blind was never broken, and data was not collected on the outcome measures.
Arm/Group | Overall Study
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Flow-mediated Dilation (FMD)
Description: Flow mediated vasodilation of the brachial artery is a measure of endothelium-dependent vasodilation. Higher flow-mediated dilation (FMD), measured as the diameter of the brachial artery in millimeters, and reported as percent change after a flow stimulus compered to basal measurement, is better, indicative of better endothelial function.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Arm/Group | Overall Study
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Change in Maximal Treadmill Walking Time
Description: Maximal treadmill walking time is measured in minutes or seconds. Higher values indicate a better outcome.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Arm/Group | Overall Study
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Change in Pain-free Treadmill Walking Time
Description: Pain-free treadmill walking time is measured in minutes or seconds. Higher values indicate a better outcome.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Arm/Group | Overall Study
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Change in Oxygen Consumption
Description: Oxygen consumption is measured in ml/kg/min. Higher values indicate better outcomes.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Arm/Group | Overall Study
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Change in Six Minute Walk Test
Description: The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes.The 6 MWT is measured in meters, and higher values indicate better outcomes.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Arm/Group | Overall Study
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: "0" Total Number of Participants at Risk (e.g., "All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events) were not monitored/assessed.
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes